CLINICAL TRIAL: NCT00609856
Title: Differences in Metabolic and Cardiovascular Effects of Pioglitazone vs. Insulin Glargine in the Treatment of Secondary Drug Failure in Type 2 Diabetes
Brief Title: Pioglitazone vs. Insulin Glargine in the Treatment of Secondary Drug Failure in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Skane University Hospital (Other)
Collaborators: Medical Research Council (Other Government); Skane County Council Research & Development Foundation (Unknown)
Responsible Party: Mozhgan Dorkhan/MD, Department of Clinical Sciences, Division of Diabetes & Endocrinology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 111/2004; 0
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2008-02-07 (Estimated); Status verified 2008-01

CONDITIONS: Type 2 Diabetes; Secondary Drug Failure
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Pioglitazone
  Interventions: Drug: pioglitazone
- 2 (Active Comparator): Insulin glargine
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: pioglitazone — tablet, 30 mg, once daily, 26 weeks
  Other Names: Actos
  Arms: 1
Drug: insulin glargine — subcutaneous injection, start dose 6-10 units, once daily, 26 weeks
  Other Names: Lantus
  Arms: 2

SUMMARY:
Pioglitazone and insulin glargine are equally effective in achieving glycemic control in secondary drug failure of type 2 diabetes but the mechanisms of actions are different.

DETAILED DESCRIPTION:
The present study was undertaken to assess differences in how insulin glargine vs. pioglitazone affect:

* Beta-cell function as measured by proinsulin/insulin, homeostasis model assessment for insulin secretion (HOMA β-cell) and glucagon stimulated C-peptide test
* Insulin sensitivity as measured by adiponectin, homeostasis model assessment for insulin resistance (HOMA-IR) and insulin tolerance test and
* Surrogate markers of cardiovascular disease as measured by BNP, NT-pro BNP and plasma lipid profile as add-on therapy in patients with T2D and secondary drug failure. The patients' satisfaction with each treatment was also surveyed.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* inadequately controlled on 50% of maximal-dose of an insulin secretagogue and metformin

Exclusion Criteria:

* heart failure (NYHA II-IV)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Effect of pioglitazone vs. insulin glargine on beta-cell function and insulin sensitivity | 26 weeks

SECONDARY OUTCOMES:
Effect of pioglitazone vs. insulin glargine on BNP | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Leif Groop, Professor, Study Director — Department of Clinical Sciences, Division of Diabetes & Endocrinology, Lund University, Malmö University Hospital, Sweden
Locations (1):
- Malmö University Hospital, Malmo, Sweden